CLINICAL TRIAL: NCT04807348
Title: A Randomised Double-blind Placebo Parallel Controlled Phase Ⅲ Clinical Study to Evaluate the Efficacy and Safety of Chiglitazar Added to Metformin in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy (RECAM)
Brief Title: Chiglitazar Added to Metformin for Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGZ303
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — chiglitazar; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chiglitazar sodium 32mg QD+metformin (Experimental): Chiglitazar 32mg qd+metformin
  Interventions: Drug: Chiglitazar 32mg; Drug: Metformin Hydrochloride
- Chiglitazar sodium 48 mg QD+metformin (Experimental): Chiglitazar 48 mg qd+metformin
  Interventions: Drug: Chiglitazar 48mg; Drug: Metformin Hydrochloride
- placebo+metformin (Placebo Comparator): placebo+metformin
  Interventions: Drug: Placebo; Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Chiglitazar 32mg — Administrated once daily
  Other Names: Bilessglu; CS038
  Arms: Chiglitazar sodium 32mg QD+metformin
Drug: Chiglitazar 48mg — Administrated once daily
  Other Names: Bilessglu; CS038
  Arms: Chiglitazar sodium 48 mg QD+metformin
Drug: Placebo — Placebo of Chiglitazar
  Other Names: Chiglitazar simulator
  Arms: placebo+metformin
Drug: Metformin Hydrochloride — most tolerable dose
  Other Names: Glucophage

SUMMARY:
The purpose of the trial is to evaluate the effect of Chiglitazar added to metformin to type 2 diabetes Inadequately controlled with metformin Monotherapy.

DETAILED DESCRIPTION:
This clinical trial is a multi-center, randomized, double-blind, placebo parallel control design, and uses superiority test to determine whether the experimental group is superior to the control group in terms of main efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. ) Provide a signed and dated informed consent form;
2. ) Men and women aged ≥ 18 years and ≤ 75 years;
3. ) According to the World Health Organization ( the WHO ) 1999 criteria for the diagnosis of type 2 diabetes;
4. ) After metformin stable dose monotherapy (≥1500 mg/day or maximum tolerated dose, but the maximum tolerated dose not < l000 mg/day) for at least 8 weeks;
5. ) The local HbA1c value during the screening period: 7.5% ≤ HbA1c ≤ 11% ;
6. ) The HbA1c value of the central laboratory before randomization: 7.0% ≤ HbA1c ≤ 10.5% ;
7. ) BMI ≥ 18.5 kg/m2 and ≤ 35 kg/m 2 ;
8. ) Fasting C- peptide ≥ 0.5 nmol/L ;
9. ) Women of Childbearing Potential ( WOCBP ) should take reliable contraceptive measures at least 1 month before the screening, during the entire trial, and within 3 months after completing the trial; male subjects should take reliable contraceptive measures to avoid making their sexual partners to pregnant during the entire trial and within 3 months after the trial.

Exclusion Criteria:

1. ) Type 1 diabetes;
2. ) Pregnancy or lactation;
3. ) The New York Heart Association (NYHA ) defines congestive heart failure as grade III or IV ;
4. ) Significant history of cardiovascular and cerebrovascular diseases within 6 months before screening, defined as myocardial infarction, coronary artery bypass graft or angioplasty, valvular disease or repair, unstable angina, transient brain Ischemic attack, or cerebrovascular accident;
5. ) Suffered from malignant tumors (except cured basal cell carcinoma) within 5 years before screening;
6. ) Edema of lower limbs or edema of the whole body;
7. ) Moderate to severe renal insufficiency [ Calculated eGFR<60 ml/ ( min*1.73m2 ) using CKD - EPI formula ];
8. ) urinary albumin-to-creatinine ratio of > 300 mg /g;
9. ) Triglyceride> 5.6 mmol /L;
10. ) Active liver disease and /or obvious liver function abnormalities, defined as AST>2.5 times the upper limit of normal value and/or ALT>2.5 times the upper limit of normal value and/or total bilirubin >1.5 times the normal value Upper limit
11. ) Clinically significant arrhythmias in the electrocardiogram examination and treatment or intervention are required. The investigator judges that it is not suitable to participate in this clinical trial;
12. ) Human immunodeficiency virus (HIV) antibody-positive; Treponema pallidum antibody positive; positive hepatitis B surface antigen and HBV DNA quantification values were higher than the upper; HCV antibodies and HCV RNA quantification values were higher than the upper ;
13. ) History of illegal drug abuse within 12 months before screening ;
14. ) Participated in other clinical trials within 90 days before screening ;
15. ) Donated whole blood, plasma, or platelets within 3 months before screening.
16. ) Before randomization, the investigator judged that the subjects had poor compliance with the study protocol or drug treatment, defined as the subjects taking less than 80% or more than 120% of the prescribed dose of chiglitazar/ placebo or metformin;
17. ) The investigator judged that it is not suitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
percentage of HbA1c change from baseline | 24 weeks
  central lab test

SECONDARY OUTCOMES:
Changes in blood fasting plasma glucose level from baseline | 12 and 24 weeks
  central lab test
Changes of HOMA-the IR value from baseline | 12 and 24 weeks
  model calculated
Changes of blood lipids level from baseline | 12 and 24 weeks
  includeing TC, LDL-C, HDL-C, VLDL-C, non-HDL-C, TG, FFA, ApoA1, ApoB
percentage of AEs | 28 weeks
  safety
number of participants with lab abnormality | 24 weeks
  number or rate of founds in lab tests

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Prof., Principal Investigator — Peking University People's Hospital
Locations (50):
- China (50):
  - Hefei Second People's Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Chang Gung Memorial Hospital, Beijing, Beijing Municipality
  - Beijing University First Hospital, Beijing, Beijing Municipality
  - Chinese People's Liberation Army Rocket Army Characteristic Medical Center, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Three Gorges Hospital Affiliated to Chongqing University, Wanzhou, Chongqing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Union Shenzhen Hospital of Huazhong University of Science and Technology, Shenzhen, Guangdong
  - Harrison International Peace Hospital, Hengshui, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The Third People's Hospital of Luoyang City, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The First People's Hospital of Chenzhou City, Chenzhou, Hunan
  - Yueyang Second People's Hospital, Yueyang, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Inner Mongolia Baotou Steel Hospital, Baotou, Inner Mongolia
  - The First People's Hospital of Huai'an, Huaian, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Yifu Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Harbin, Jilin
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Jilin
  - The Second Hospital of Jilin University, Harbin, Jilin
  - Panjin Liaoyou Baoshihua Hospital, Panjin, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical College, Shandong Province, Jining, Shandong
  - Qingdao University Hospital, Qingdao, Shandong
  - Gongli Hospital, Pudong New Area, Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Minhang District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Shanghai, Shanghai Municipality
  - Shanghai Seventh People's Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Central Hospital of Yuncheng City, Shanxi Province, Yuncheng, Shanxi
  - Tangshan Workers' Hospital, Tangshan, Tianjin Municipality
  - Huzhou Central Hospital, Huzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ji L, Song W, Fang H, Li W, Geng J, Wang Y, Guo L, Cai H, Yang T, Li H, Yang G, Li Q, Liu K, Li S, Liu Y, Shi F, Li X, Gao X, Tian H, Ji Q, Su Q, Zhou Z, Wang W, Zhou Z, Li X, Xu Y, Ning Z, Cao H, Pan D, Yao H, Lu X, Jia W. Efficacy and safety of chiglitazar, a novel peroxisome proliferator-activated receptor pan-agonist, in patients with type 2 diabetes: a randomized, double-blind, placebo-controlled, phase 3 trial (CMAP). Sci Bull (Beijing). 2021 Aug 15;66(15):1571-1580. doi: 10.1016/j.scib.2021.03.019. Epub 2021 Mar 23. PMID 36654286
- [Result] Jia W, Ma J, Miao H, Wang C, Wang X, Li Q, Lu W, Yang J, Zhang L, Yang J, Wang G, Zhang X, Zhang M, Sun L, Yu X, Du J, Shi B, Xiao C, Zhu D, Liu H, Zhong L, Xu C, Xu Q, Liang G, Zhang Y, Li G, Gu M, Liu J, Yuan G, Yan Z, Yan D, Ye S, Zhang F, Ning Z, Cao H, Pan D, Yao H, Lu X, Ji L. Chiglitazar monotherapy with sitagliptin as an active comparator in patients with type 2 diabetes: a randomized, double-blind, phase 3 trial (CMAS). Sci Bull (Beijing). 2021 Aug 15;66(15):1581-1590. doi: 10.1016/j.scib.2021.02.027. Epub 2021 Feb 16. PMID 36654287
- [Derived] Gao L, Ji L, Yan X, Cheng Z, Zhang X, Sun W, Ma J, Song W, Liu Y, Lin X, Pang W, Cao H, Chen B, Li Z, Lu X; RECAM Study Group. Efficacy and safety of chiglitazar add-on to metformin in type 2 diabetes mellitus (RECAM study). Diabetes Obes Metab. 2025 Nov;27(11):6243-6253. doi: 10.1111/dom.70009. Epub 2025 Aug 22. PMID 40842343